CLINICAL TRIAL: NCT02777671
Title: Effect of Eslicarbazepine Acetate on the Pharmacokinetics of Gliclazide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-126
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Period 1 - BIA 2-093 + Gliclazide Period 2 - Gliclazide
  Interventions: Drug: BIA 2-093; Drug: Gliclazide
- Group B (Experimental): Period 1 - Gliclazide Period 2 - BIA 2-093 + Gliclazide
  Interventions: Drug: BIA 2-093; Drug: Gliclazide

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate
Drug: Gliclazide — tablets containing gliclazide 80 mg (Diamicron® 80 mg)

SUMMARY:
Single centre, randomised, open-label, two-way crossover study to investigate whether multiple-dose administration of eslicarbazepine acetate (ESL, BIA 2-093) affects the pharmacokinetics of gliclazide.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for the study if they fulfilled all of the following inclusion criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening
* Clinical laboratory test results clinically acceptable at screening and admission to each treatment period.
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Non-smokers or who smoke ≤ 10 cigarettes or equivalent per day.
* Able and willing to give written informed consent.
* (If female) Not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier or intrauterine device.
* (If female) Negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

Subjects were not eligible for the study if they fulfilled any of the following exclusion criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Clinically relevant surgical history.
* History of relevant atopy or drug hypersensitivity.
* History of alcoholism or drug abuse.
* Consumed more than 14 units of alcohol a week.
* Significant infection or known inflammatory process at screening or admission to each treatment period.
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period.
* Used medicines within 2 weeks of admission to first period that may affect the safety or other study assessments, in the investigator's opinion.
* Used any investigational drug or participated in any clinical trial within 6 months prior to screening.
* Participated in more than 2 clinical trials within the 12 months prior to screening.
* Donated or received any blood or blood products within the 3 months prior to screening.
* Vegetarians, vegans or with medical dietary restrictions.
* Could not communicate reliably with the investigator.
* Unlikely to co-operate with the requirements of the study.
* Unwilling or unable to give written informed consent.
* (If female) Pregnant or breast-feeding.
* (If female) Of childbearing potential and she did not use an approved effective contraceptive method (double-barrier or intra-uterine device) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cmax | before the gliclazide dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h post-gliclazide dose
  Maximum plasma concentration (Cmax) of Gliclazide following a single oral dose of 80 mg administered alone
Tmax | before the gliclazide dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h post-gliclazide dose
  Time to maximum observed concentration (Tmax) of Gliclazide following a single oral dose of 80 mg administered alone
AUC0-12 | before the gliclazide dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h post-gliclazide dose
  Area under the plasma concentration-time curve over 12 hours (AUC0-12) of Gliclazide following a single oral dose of 80 mg administered alone
AUC0-∞ | before the gliclazide dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h post-gliclazide dose
  Area under the concentration-time curve from time zero up to infinity with extrapolation of the terminal phase (AUC0-∞) of Gliclazide following a single oral dose of 80 mg administered alone

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit, S. Mamede Do Coronado, Portugal